CLINICAL TRIAL: NCT03090399
Title: Effects of the Goal-directed Fluid Therapy on ASA 1 Patients Scheduled for Intensive Debulking Surgery
Brief Title: Fluid ORiented Therapy for yoUNg Asa 1patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.Andrea Russo, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORTUNA study
Record Dates: First submitted 2017-01-13; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Hemodynamics
Keywords: Goal Directed Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): patients in which standard fluid administration was applied
- case group (Active Comparator): patients in which fluids were administered according to FloTrac parameters
  Interventions: Device: FloTrac

INTERVENTIONS:
Device: FloTrac — For patients belonging to case group a Pulse Contour Analysis was adopted for optimize fluid administration
  Arms: case group

SUMMARY:
In this retrospective analysis investigators will study the effects of using a minimally invasive hemodynamic monitoring (FloTrac-Edwards) on postoperative outcomes. Participants will compare a control group to a case group; in both groups ASA 1 patients suffering from advanced ovarian cancer underwent radical cytoreductive surgery. In case group hemodynamic was managed by using the FloTrac system; in the control group a standard hemodynamic monitoring was used.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1

Exclusion Criteria:

* cardiac diseases
* pulmonary diseases
* renal diseases
* metabolic disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
prevalence of complications | up to 30 days

SECONDARY OUTCOMES:
days of hospitalization | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea MD Russo, Principal Investigator — Department of Anesthesiology

IPD SHARING:
Plan to Share IPD: Yes